CLINICAL TRIAL: NCT04857021
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Clinical Study to Investigate the Sleep Quality Enhancing Effect and Safety of Lactobacillus-fermented GABA in Subjects With Mild, Transient Sleep Disorder
Brief Title: Clinical Study to Investigate the Sleep Quality Enhancing Effect of GABA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AP-PV-2018-01
Record Dates: First submitted 2021-04-14; First posted 2021-04-23 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-06

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias | interventions — gamma-Aminobutyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GABA (Active Comparator): Take GABA capsule once daily before sleep for 14 days.
  Interventions: Dietary Supplement: GABA
- Placebo (Placebo Comparator): Take placebo capsule once daily before sleep for 14 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GABA — oral administration of GABA capsule once daily before sleep
  Other Names: Lactobacillus brevis-fermented
  Arms: GABA
Dietary Supplement: Placebo — oral administration of placebo capsule once daily before sleep
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of dietary supplement GABA in subjects with mild, transient sleep disorder.

DETAILED DESCRIPTION:
The subjects will take GABA or placebo capsule once daily before sleep for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects older than 19 years old
* Who is experiencing mild, transient sleep disturbance (pittsburgh sleep quality index ≥ 5, Insomnia Severity Index ≥ 8)
* Who voluntarily agreed to participate in the study and signed an informed consent form.

Exclusion Criteria:

* Who is suffering from severe sleep disorder including sleep disorders due to psychological or neurologic causes.
* Who has used sleeping pills or sleep related dietary supplements within 4 weeks before study participation
* Who is suffering from obstructive sleep apnea.
* Who has used or is expected to inevitably use prohibited concomitant medications during the study.
* Women who is pregnant /breast-feeding, or who has childbearing potential and does not use available contraceptives.
* Who has dosed other study medications within 30 days before screening.
* Who is determined ineligible for study participation by investigators for any other reasons.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-14 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Change of total sleep time of polysomnography | Baseline, Week 2
  total sleep time(minutes)
Change of sleep latency of polysomnography | Baseline, Week 2
  sleep latency(minutes)
Change of sleep efficiency of polysomnography | Baseline, Week 2
  sleep efficiency(percent)
Change of NonREM stage3 of polysomnography | Baseline, Week 2
  NonREM stage3(mintues)
Change of total wake time of polysomnography | Baseline, Week 2
  total wake time(mintues)
Change of wake after sleep onset of polysomnography | Baseline, Week 2
  wake after sleep onset(mintues)

SECONDARY OUTCOMES:
Change of Pittsburgh Sleep Quality Index | Baseline, Week 2
  Change of Pittsburgh Sleep Quality Index(0-21), higher score means worse outcome
Change of Insomnia Severity Index | Baseline, Week 2
  Change of Insomnia Severity Index(0-28), higher score means worse outcome
Change of Epworth sleepiness scale | Baseline, Week 2
  Change of Epworth sleepiness scale(0-24), higher score means worse outcome
Change of Fatigue Severity Scale | Baseline, Week 2
  Change of Fatigue Severity Scale(9-63), higher score means worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Kyunghee University Hospital at Gangdong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No